CLINICAL TRIAL: NCT07042230
Title: Proprioceptive Neuromuscular Facilitation And Passive Vertebral Mobilization For Neck Disability In Patients With Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Umaima Naeem, Physiotherapist, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/506/08/24
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain; Neck Pain Musculoskeletal; Mechanical Neck Pain; Proprioceptive Neuromuscular Facilitation; Mobilization
Keywords: Articular; Cervical Vertebrae; Manual Therapy; Neck Pain; Proprioception; Range of Motion
MeSH Terms: conditions — Neck Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation (PNF) (Experimental): Participants in this arm received Proprioceptive Neuromuscular Facilitation (PNF) techniques aimed at improving neck mobility, pain, and function. The intervention included rhythmic initiation, dynamic reversals, and contract-relax techniques performed across four cranio-cervical diagonal movement patterns (e.g., extension with left rotation, flexion with right rotation). Each session lasted 15-30 minutes and was delivered three times per week for four weeks. Techniques were progressed based on patient tolerance, with repetitions increased in the third and fourth weeks. All sessions were administered by licensed physiotherapists following standardized protocols.
  Interventions: Other: Proprioceptive Neuromuscular Facilitation (PNF)
- Passive Vertebral Mobilization (PVM) (Experimental): Participants in this arm received Maitland-based Passive Vertebral Mobilization (PVM) techniques targeting cervical vertebrae to improve joint mobility and reduce neck pain. Mobilizations were applied in prone lying using posteroanterior central and unilateral glides. Treatment began with Grades I-II oscillatory mobilizations in Weeks 1-2, progressing to Grades III-IV in Weeks 3-4, based on patient response and tolerance. Each session lasted 15-20 minutes and was conducted three times per week for four weeks. Interventions were performed by trained physiotherapists using standardized procedures.
  Interventions: Other: Passive Vertebral Mobilization (PVM)

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation (PNF) — Proprioceptive Neuromuscular Facilitation (PNF) techniques were applied to the cervical region using rhythmic initiation, dynamic reversals, and contract-relax methods. Movements followed diagonal cranio-cervical patterns including flexion/extension with rotational components. Each session lasted 15-30 minutes, delivered three times per week for four weeks. Repetitions and sets were progressively increased based on patient tolerance. The goal was to enhance neuromuscular coordination, improve cervical range of motion, and reduce pain through active facilitation techniques.
  Other Names: PNF Stretching; PNF Cervical Patterns
  Arms: Proprioceptive Neuromuscular Facilitation (PNF)
Other: Passive Vertebral Mobilization (PVM) — Passive Vertebral Mobilization (PVM) was administered using Maitland mobilization techniques applied to the cervical spine. Posteroanterior central and unilateral glides were performed with the participant in a prone position. Mobilizations started with Grades I-II during Weeks 1-2 and progressed to Grades III-IV in Weeks 3-4, depending on patient response. Each session lasted 15-20 minutes and was conducted three times weekly over four weeks. This passive manual therapy aimed to improve joint mobility, reduce muscle stiffness, and alleviate mechanical neck pain.
  Other Names: Cervical Maitland Mobilization; Spinal Mobilization Techniques
  Arms: Passive Vertebral Mobilization (PVM)

SUMMARY:
Mechanical neck pain is a common musculoskeletal condition that affects many people, especially those with poor posture or repetitive neck movements. It can cause discomfort, reduce the ability to move the neck, and affect daily functioning. This study aimed to compare the effects of two physiotherapy treatments-Proprioceptive Neuromuscular Facilitation (PNF) and Passive Vertebral Mobilization (PVM)-on neck pain, disability, and movement.

This randomized controlled trial was conducted at the University of Lahore Teaching Hospital over nine months. A total of 62 participants, aged 18 to 35 years, who had mechanical neck pain for at least four weeks, were recruited and randomly assigned to one of two groups: Group A received PNF, while Group B received PVM. Both treatments were delivered by physiotherapists three times per week for four weeks.

PNF is an active therapy that involves specific movement patterns to improve muscle coordination and flexibility. PVM is a passive manual therapy technique where the therapist gently moves the neck vertebrae to improve joint mobility and reduce pain.

Outcomes were measured using the Neck Disability Index (NDI), the Numeric Pain Rating Scale (NPRS), and measurements of neck movement (Active Cervical Range of Motion, or ACROM) at the start of the study, at two weeks, and at the end of the four-week treatment. The study was single-blinded-meaning the person assessing the outcomes did not know which treatment the patient received.

The results showed that both treatments significantly improved pain, movement, and function. However, the group that received PNF showed slightly greater reduction in pain scores by the end of the treatment. There were no significant differences between the groups in terms of disability or movement range.

This study concluded that both PNF and PVM are beneficial treatments for mechanical neck pain. PNF may offer slightly faster pain relief, while both interventions are effective at improving mobility and reducing neck-related disability. These findings can help guide physiotherapists and patients in choosing suitable treatment options for neck pain.

DETAILED DESCRIPTION:
Mechanical neck pain is a common musculoskeletal condition often caused by poor posture, repetitive stress, or mechanical strain involving cervical joints, ligaments, and muscles. It is typically localized and not associated with radiating symptoms. This condition leads to functional disability, reduced cervical range of motion (ROM), and increased pain, significantly affecting individuals' quality of life and work productivity. While various physiotherapeutic approaches are employed in its management, the comparative efficacy of Proprioceptive Neuromuscular Facilitation (PNF) and Passive Vertebral Mobilization (PVM) remains inadequately explored in controlled settings.

This randomized controlled trial aimed to evaluate and compare the effectiveness of PNF and PVM techniques in improving neck-related disability, reducing pain, and enhancing active cervical ROM in individuals diagnosed with mechanical neck pain. The study was conducted at the University of Lahore Teaching Hospital and followed ethical approval and informed consent protocols. The trial design was single-blinded, with the assessor unaware of group allocation.

A total of 62 participants aged 18-35 years with clinically diagnosed mechanical neck pain of at least 4 weeks duration were included using purposive sampling. Participants were randomly allocated (via lottery method) into two equal groups (n = 31 per group): Group A received PNF techniques, and Group B received Maitland-based passive vertebral mobilization.

Group A (PNF) intervention involved rhythmic initiation, dynamic reversals, and contract-relax patterns performed across diagonal cranio-cervical movement patterns. Group B (PVM) received graded Maitland mobilizations (Grades I-IV) targeting the cervical vertebrae. Both groups received physiotherapy three times per week for four consecutive weeks. Each treatment session lasted 15-30 minutes.

Outcome measures were recorded at baseline, week 2, and week 4 and included:

Neck Disability Index (NDI): to assess functional limitation

Numeric Pain Rating Scale (NPRS): to measure subjective pain intensity

Active Cervical Range of Motion (ACROM): measured using a goniometer

Statistical analysis using SPSS Version 24 revealed that both groups experienced statistically significant improvements over time in all outcome measures:

NDI (F = 355.163, p < .001)

NPRS (F = 544.090, p < .001)

ACROM (F = 33.413, p < .001)

Between-group comparisons showed no significant difference for NDI (p = .769) or ACROM (p = .987). However, PNF demonstrated significantly greater pain reduction at baseline (p = .039) and at week four (p = .043), suggesting superior short-term analgesic effects.

This trial demonstrated that both PNF and PVM are effective in reducing neck disability and improving cervical mobility and pain. PNF may offer enhanced short-term pain relief due to its neuromuscular activation mechanisms, while PVM remains an effective passive intervention for joint mobilization.

The study's findings provide clinicians with evidence supporting both interventions, allowing treatment selection based on individual patient presentation, therapist skill, and rehabilitation goals. Future studies with larger samples and longer follow-up periods are recommended to assess long-term efficacy, retention of benefits, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 35 years were included in the study (Ashfaq et al., 2022).
* Participants diagnosed with pain localized in the neck region for at least 4 weeks were included.
* Participants diagnosed with no radiating pain beyond the shoulder or fingers were included (Cohen, 2015).
* Participants diagnosed with no identified neurological deficits were included.
* Participants having no history of major trauma or surgery to the cervical spine were included (Rodríguez-Huguet et al., 2020).

Exclusion Criteria:

* Participants who were diagnosed with ankylosing spondylitis, rheumatoid arthritis, fracture of spine, cancer or congenital anomaly of the cervical spine, positive neurological findings (Ashfaq et al., 2022).
* Patients with any other contraindication to manual therapy (Ashfaq et al., 2022).
* Neurological conditions affecting the cervical spine.
* Uncontrolled dizziness or vertigo (Cohen, 2015).
* Known malignancy or any pregnancy (Cohen, 2015).
* Current use of medications that could affect pain perception (e.g., opioids, high-dose antidepressants) (Rodríguez-Huguet et al., 2020)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Neck Disability | Baseline, Week 2, and Week 4
  The Neck Disability Index (NDI) is a validated, self-reported questionnaire that assesses disability related to neck pain. It contains 10 items, each scored from 0 to 5, with higher scores indicating greater disability. The total score ranges from 0 to 50 and is converted into a percentage. This outcome will assess improvement in neck-related function and disability following 4 weeks of intervention with either PNF or PVM.

SECONDARY OUTCOMES:
Cervical Pain | Baseline, Week 2, and Week 4
  The Numeric Pain Rating Scale (NPRS) is an 11-point self-reported scale ranging from 0 ("no pain") to 10 ("worst imaginable pain"). It is used to quantify the patient's subjective pain intensity. Changes in NPRS scores will be recorded to assess the effectiveness of the interventions in reducing neck pain.
Active Cervical Range of Motion (ACROM) | Baseline, Week 2, and Week 4
  ACROM will be measured using a universal goniometer in degrees across cervical flexion, extension, lateral flexion, and rotation. This measure will assess the improvement in neck mobility and functional range following intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No